CLINICAL TRIAL: NCT00890110
Title: Phase1/2 Study of Vaccination With DNP Modified Autologous Renal Cell Carcinoma in Combination With Sunitinib in Stage 4 RCC
Brief Title: Autologous Vaccination of Stage 4 Renal Cell Carcinoma Combined With Sunitinib
Acronym: rcc
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Hovav Nechushtan - MD PhD attending Physician Oncology department, Hadassah Ein Kerem Medical center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCC- vac-sut-1
Record Dates: First submitted 2009-04-26; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Renal Cell Cancer
Keywords: Renal cell cancer; sunitinib; autologous vaccine; metastatic RCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologus vaccination with suntinib (Experimental): Combination of autologous dnp irradiated modified cells with sunitinib treatments
  Interventions: Biological: Autologous renal cell vaccine based on DNP modified cells

INTERVENTIONS:
Biological: Autologous renal cell vaccine based on DNP modified cells — Primary or metastatic tumor resected in an Israeli hospital will be used to derive autologous cell lines used for vaccinations following DNP modifications in combination with the regular Sunitinib treatments. Immunological and clinical followup of the patients will be performed
  Other Names: autologous vaccine for rcc tumors with sunitinib

SUMMARY:
While different lines of evidence support the notion that renal cell cancer is amenable for immunologic vaccination, up to now the clinical benefit associated with vaccines has been limited. One reason being probably the whole immunological state of the patients with RCC in which the tumor releases various substances promoting tolerance of the immune system towards the carcinoma. Recent data demonstrates that sunitinib has effects on the immune system which might enhance effectivity of anti tumor vaccines.

Since in kidney cancer it is quite common to resect primary tumor when there are few metastasis or or metastatic tumor resected (if there are few metastasis), the investigators plan to use these tumor source to grow autologous carcinoma cell lines and use a method used world wide for many years and in our institution for over a decade to modify these cells by dinitro phenol and use irradiated cell for patients vaccination in combination with sunitinib treatments.

The investigators will monitor clinical and immunological parameters in these patients.

DETAILED DESCRIPTION:
Background: Renal cell carcinoma (RCC) constitutes around 3% of all solid tumors and cure for metastatic sidease is reported for less than 5% of patients. Together with melanoma it is considered the most immune responsive tumor, moreover it is a common practice to resect primary tumor or large metastasis even in the metastatic settings. Antiangiogenesis treatments are currently the favored antitumor drugs, however their use has rarely resulted in complete response/ cure. Recently it has been demonstrated that these drugs can elicit a shift in the immune environment in RCC patients (improved T1 responses reduced Treg responses).Our department has experience in the treatment 200 melanoma patients with cellular vaccination and in the preparation of primary tumor cell lines from various tumors including RCC. Interestingly , immune modulators such as antiCTLA-4 Ab have demonstrated impressive activity in patients previously vaccinated with cellular vaccinations.

Working hypothesis: Vaccination with autologous cellular vaccines of RCC patients will induce clinical and immunological responses and help in formulation of better combined vaccination strategies in this cancer. Our aims are: 1) Growth and characterization of primary RCC cell lines,2)vaccination with autologous cellular vaccines in combination with sunitinib. 3) Clinical and immunologic characterizations for derivation of prognostic and predictive factors.

Methods: primary or metastatic tumor resected in one of several Israeli hospitals will be used to derive autologous cell lines used for vaccinations following DNP modifications in combination with the regular Sunitinib treatments. Immunological and clinical followup of the patients will be performed and primary cell lines will be grown for further in-vitro testing including possible future use for allogeneic vaccines. Expected result Good safety profile combined with significant clinical and immunological responses are expected.

Importance: This research might result in clinical benefit to the treated patients and will be important in the formulation of effective immune strategies in kidney cancer.

Probable implications to Medicine: RCC vaccine in combination with other therapies has the potential to lead to longer survival and even cure the proposed study will help in the formulation of such a vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic renal cell cancer
* Primary/metastatic tumor for which resection seems of potential clinical benefit and fresh tissue can be obtained
* Patients for whom treatment with Sunitinib is the preferred clinical therapy
* Ecog <2
* Willingness to participate in the trial and contribute small amounts ( up to 100cc for all the trial) of blood for immunological monitoring
* No concurrent active cancers ( excluding cancers which are not life threatening such as localized treated low grade prostate cancer,skin cancer etc)

Exclusion Criteria:

* Age under 70
* Life expectancy less than 3 months
* Large tumor burden at multiple organs

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
immunological response to therapy | two years

SECONDARY OUTCOMES:
patients progression free survival | until end of 2011
dermatologic and allergic reactions to vaccine injections | during active treatments period

CONTACTS AND LOCATIONS:
Overall Officials: Hovav Nechushtan, MD PHD, Principal Investigator — Hadassah Medical Organization

REFERENCES:
- [Background] Lotem M, Shiloni E, Pappo I, Drize O, Hamburger T, Weitzen R, Isacson R, Kaduri L, Merims S, Frankenburg S, Peretz T. Interleukin-2 improves tumour response to DNP-modified autologous vaccine for the treatment of metastatic malignant melanoma. Br J Cancer. 2004 Feb 23;90(4):773-80. doi: 10.1038/sj.bjc.6601563. PMID 14970852
- [Background] Ko JS, Zea AH, Rini BI, Ireland JL, Elson P, Cohen P, Golshayan A, Rayman PA, Wood L, Garcia J, Dreicer R, Bukowski R, Finke JH. Sunitinib mediates reversal of myeloid-derived suppressor cell accumulation in renal cell carcinoma patients. Clin Cancer Res. 2009 Mar 15;15(6):2148-57. doi: 10.1158/1078-0432.CCR-08-1332. Epub 2009 Mar 10. PMID 19276286
- [Background] Hutson TE, Figlin RA, Kuhn JG, Motzer RJ. Targeted therapies for metastatic renal cell carcinoma: an overview of toxicity and dosing strategies. Oncologist. 2008 Oct;13(10):1084-96. doi: 10.1634/theoncologist.2008-0120. Epub 2008 Oct 6. PMID 18838439
- See also: just a sight describing all the publication in which the principle investigator had a contribution — http://www.biomedexperts.com/Profile.bme/1008720/Hovav_Nechustan